CLINICAL TRIAL: NCT05156749
Title: Unterarm-Combicast Versus Oberarm-Combicast Bei Gelenknahen Distalen (Salter Harris I/II) Radius- Und Vorderarmfrakturen Im Kindesalter
Brief Title: Short and Long-arm Fiberglass Cast Immobilization for Distal Salter Harris I and II Forearm Fractures in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UChildrenZurich_salter harris
Record Dates: First submitted 2021-11-29; First posted 2021-12-14 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Fracture Forearm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- short-arm fiberglass cast (Experimental): salter harris fractures of the distal radius/forearm in children are usually treated with fiberglass long-arm casts. The investigators were able to demonstrate that in distal metaphyseal forearm fracture, treatment with a short-arm cast is not inferior to a long-arm cast.
  Patients are going to receive a short-arm cast for fracture treatment.
  Interventions: Device: short-arm fiberglass cast
- long-arm fiberglass cast (Active Comparator): salter harris fractures of the distal radius/forearm in children are usually treated with a fiberglass long-arm cast.
  Patients are going to receive a long-arm cast for fracture treatment.
  Interventions: Device: long-arm fiberglass cast

INTERVENTIONS:
Device: short-arm fiberglass cast — fracture stabilization of salter harris I/II fractures with a fiberglass short-arm cast
  Arms: short-arm fiberglass cast
Device: long-arm fiberglass cast — fracture stabilization of salter harris I/II fractures with a fiberglass long-arm cast
  Arms: long-arm fiberglass cast

SUMMARY:
The aim of this study is to investigate whether short-arm fiberglass cast (SAC) immobilization provides fracture stabilization comparable to that of long-arm cast (LAC) treatment of displaced and non-displaced distal Salter Harris I/II forearm fractures in paediatric patients.

DETAILED DESCRIPTION:
The patients are allocated randomly into the two groups(short-arm cast, long-arm cast). After confirming study participation, patients draw a sealed envelope enclosing a numbered card, which assignes them to one group or other. After choosing the envelope, neither the ED staff nor the parents and their childrenare blinded for the treatment groups. However, the data are going to be analyzed under blinded conditions

ELIGIBILITY:
Inclusion Criteria:

* Salter Harris I or II fracture of the distal radius or a forearm fracture
* informed consent

Exclusion Criteria:

* open/instable/intraarticular fracture
* age <4 years or > 16years
* no informed consent

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of fracture displacement | in the first four weeks after trauma
  difference in fracture angulation values either at pre-treatment or during follow-up between the two groups (short-arm cast; long-arm cast)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Seiler, PD, Study Chair — University Children's Hospital, Zurich
Locations (1):
- University Children's Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No